CLINICAL TRIAL: NCT03517332
Title: Circulating Tumor DNA Exposure in Peripheral Blood Using a Novel Process: A Feasibility Study
Brief Title: Circulating Tumor DNA Exposure in Peripheral Blood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Quantgene Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: QG01012015
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer; Pancreatic Adenocarcinoma; Gastric Cancer; Hepatocellular Carcinoma; Non-small Cell Lung Cancer; Bladder Cancer; Melanoma; Ovarian Cancer; Adrenocortical Cancer; Breast Cancer; Other Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Melanoma; Ovarian Neoplasms; Adrenal Cortex Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA in blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Have a diagnosis of a malignancy in clinical stage 0 to IV including but not limited to: colon or rectal cancer, pancreatic and gastric cancer, hepatocellular carcinoma, non-small cell lung cancer, bladder cancer, melanoma
  Subjects of cohort 1 must not:
  • Have been treated for above diagnosed malignancy
- Cohort 2: Negative cohort with subjects that have not been diagnosed with a malignancy (cohort 2).
  Subjects of cohort 2 must:
  • Meet the listed matching criteria
  Subjects of cohort 2 must not:
  • Have been diagnosed/treated for a malignancy previously

SUMMARY:
This is a prospective, multi-center, blinded feasibility study. The objective of this study is to test the feasibility of the detection of tumor DNA of a variety of tumors in peripheral blood using a novel process for the detection of circulating tumor DNA (ctDNA).

DETAILED DESCRIPTION:
This prospective, multi-center, feasibility study represents a feasibility study to determine the potential of circulating tumor DNA exposure in peripheral blood using a novel process in a sample of patients with different types of malignant organ tumors and a control cohort without malignant disease. The study applies a new process to detect ctDNA and other molecular markers in peripheral blood using: a collection of de-identified blood specimen and clinical data from up to 10,000 participants from clinical sites across the United States and Europe. Data collected will include the following: Demographics, Tumor Characteristics, Information about Treatment, Specimen Assessment, Postoperative Assessment Clinical information, and Follow-up at intermittent future time points, for up to 15 years. The study test(s) to be used in this protocol is a multiplexed primer and probe design developed, that allows detecting a wider set of mutations at a higher sensitivity then conventional sequencing-based method. This novel process is currently being investigated at Quantgene Inc.

ELIGIBILITY:
Inclusion Criteria:

* This study will include subjects that are diagnosed with a malignancy (cohort

  1) and a negative cohort with subjects that have not been diagnosed with a malignancy (cohort 2).
* Subjects of both cohorts must:

  * Be of age ≥ 18
  * Provide written consent for study participation
* Subject of cohort 1 must:

  * Have a diagnosis of a malignancy in clinical stage 0 to IV including but not limited to: colon or rectal cancer, pancreatic and gastric cancer, hepatocellular carcinoma, non-small cell lung cancer, bladder cancer, melanoma

Subjects of cohort 2 must:

• Meet the listed matching criteria

Exclusion Criteria:

* Subjects of cohort 1 must not: Have been treated for above diagnosed malignancy
* Subjects of cohort 2 must not:

  * Have been diagnosed/treated for a malignancy previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Subjects that are diagnosed with a malignancy (cohort 1)
  * Subjects that have not been diagnosed with a malignancy (cohort 2)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor DNA exposure in peripheral blood using a novel process: A feasibility study | 28 Months
  The objective of this study is to test the feasibility of the detection of tumor DNA of a variety of tumors in peripheral blood using a novel process for the detection of circulating tumor DNA (ctDNA).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Florida Hospital Celebration Health, Celebration, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Premier Surgical Oncology, Centerville, Ohio
  - Kettering Medical Center, Dayton, Ohio
- University Hospital of Geneva, Geneva, Switzerland